CLINICAL TRIAL: NCT01364402
Title: Prevention of Contrast Induced Nephropathy by Erythropoietin in Patients With Diabetes Mellitus and eGFR<60 ml/Min/1.73m2 Undergoing Percutaneous Coronary Intervention
Brief Title: Prevention of Contrast Induced Nephropathy by Erythropoietin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Dr. Shaul Atar, Western Galilee Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EPO1
Record Dates: First submitted 2011-05-24; First posted 2011-06-02 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes; Chronic Kidney Insufficiency
Keywords: scheduled for PCI
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — epoetin beta; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Experimental)
  Interventions: Drug: Epoetin beta
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Epoetin beta — 50,000U intravenously
  Other Names: Epoietin beta
  Arms: Erythropoietin
Drug: Saline 0.9% — normal saline intravenously
  Other Names: Hydration
  Arms: Placebo

SUMMARY:
This ia a prospective, randomized, double blind, placebo controlled trial. patients schedule for primary PCI or elective PCI will randomly allocated to receive either a single dose of EPO (Recormon, Roche, Epoetin beta) or saline intravenously before PCI.

The investigators assume that the incidence rate of CIN will be significantly lower in the EPO group compared to placebo. In addition, EPO administration will result in a decrease of infarct size.

DETAILED DESCRIPTION:
Radiological procedures utilizing intravascular contrast media are being widely applied for both diagnostic and therapeutic purposes. This has resulted in the increasing incidence of procedure-related contrast-induced nephropathy (CIN), which was found to be associated with poor outcome including higher in-hospital mortality rates. Therefore, finding ways to prevent CIN is a valuable clinical and research goal. However, there are no current methods for efficient and cost-effective prevention CIN. Erythropoietin (EPO) has been shown to elicit tissue-protective effects in various experimental models and few clinical studies of acute kidney injury (AKI). Therefore, this prospective, randomized, double blind, placebo controlled trial aim to evaluate, for the first time, the effectiveness of EPO in the prevention of CIN after percutaneous coronary intervention (PCI).

The potential reno-protective effect of EPO is expected to reduce the incidence of the third leading cause of hospital-acquired acute kidney injury. The above together with a cardio-protective effect of EPO is expected to reduce patient's morbidity, mortality and the high health cost associated with CIN treatment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Diabetic patients.
* eGFR < 60 ml/min/1.73m2.
* Scheduled for primary or elective PCI.

Exclusion Criteria:

* Non diabetic patients.
* Patients with eGFR ≥ 60 ml/min/1.73m2.
* Chronic renal replacement therapy.
* Subject with active malignancy.
* Subject with any known history of seizure disorders.
* Subject with polycythemia.
* Uncontrolled hypertension.
* Known allergy or hypersensitivity to EPO.
* Use of EPO 1 week prior to randomization.
* Use of long acting EPO (CERA) during 1 month prior to randomization.
* Use of NAC or bicarbonate during 3 days prior to randomization.
* Contrast media exposure during the last 7 days before randomization.
* Pregnant or lactating women.
* Participation in other clinical trial.
* Refusal or inability to give informed consent due to mental or physical state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Contrast Induced Nephropathy(CIN) | 1-3 days after exposure to contrast media

SECONDARY OUTCOMES:
Enzymatic infarct size | 6h and 12 h after exposure to contrast media
  Will be measured by Troponin and CK
Hospital length of stay | participants will be followed for the duration of hospital stay, an expected average of 3 days
Renal replacement therapy | participants will be followed after PCI procedure till discharge, an expected average of 1-2 days
Hospital mortality | participants will be followed after PCI procedure till discharge, an expected average of 1-2 days

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Atar, MD, Principal Investigator — Western Galilee Hospital
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

REFERENCES:
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879